CLINICAL TRIAL: NCT00563368
Title: A Phase III, Randomized, Double-Blind, Parallel-Design Study Comparing Multiple Doses of VI-0521 to Placebo and Their Single-Agent Phentermine and Topiramate Constituents for the Treatment of Obesity in Adults
Brief Title: A Study Comparing Multiple Doses of VI-0521 With Placebo and Their Single-agent Constituents for Treatment of Obesity in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OB-301
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Topiramate; Phentermine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- VI-0521 Top (Experimental): VI-0521; high dose phentermine/topiramate
  Interventions: Drug: VI-0521
- VI-0521 Mid (Experimental): VI-0521; mid dose phentermine/topiramate
  Interventions: Drug: VI-0521
- TPM 46 (Active Comparator): mid dose topiramate
  Interventions: Drug: topiramate
- TPM 92 (Active Comparator): high dose topiramate
  Interventions: Drug: topiramate
- PHEN 7.5 (Active Comparator): mid dose phentermine
  Interventions: Drug: phentermine
- PHEN 15 (Active Comparator): high dose phentermine
  Interventions: Drug: phentermine
- Placebo (Placebo Comparator)
  Interventions: Drug: VI-0521

INTERVENTIONS:
Drug: VI-0521 — phentermine 15 mg and topiramate 92 mg, po once daily
  Arms: VI-0521 Top
Drug: VI-0521 — phentermine 7.5 mg and topiramate 46 mg, po once daily
  Arms: VI-0521 Mid
Drug: topiramate — topiramate 46 mg, po once daily
  Arms: TPM 46
Drug: topiramate — topiramate 92 mg, po once daily
  Arms: TPM 92
Drug: phentermine — phentermine 7.5 mg, po once daily
  Arms: PHEN 7.5
Drug: phentermine — phentermine 15 mg, po once daily
  Arms: PHEN 15
Drug: VI-0521 — placebo, po once daily
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of various doses of VI-0521 compared to both placebo, and the single-agent components that comprise each combination dose. This study will provide confirmatory data to demonstrate that doses of VI-0521 have efficacy that is greater than placebo and each of the single-agent components that comprise the combination dose.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or less with body mass index (BMI) between 30 and 45 kg/m2
* Informed Consent
* Females of child-bearing potential must be using adequate contraception

Exclusion Criteria:

* Stroke/myocardial infarction (MI)/unstable cardiovascular disease within 6 months
* Clinically significant renal, hepatic or psychiatric disease
* Unstable thyroid disease or replacement therapy
* Nephrolithiasis
* Obesity of known genetic or endocrine origin
* Participation in a formal weight loss program or lifestyle intervention
* Glaucoma or elevated intraocular pressure
* Pregnancy or breastfeeding
* Drug or Alcohol abuse
* Smoking cessation within previous 3 months or plans to quit smoking during study
* Eating disorders within past year
* Cholelithiasis within past 6 months
* Type 2 diabetes
* Previous bariatric surgery
* Bipolar disorder or psychosis
* Steroid hormone therapy not stable for 3 months
* Systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Peterson, Study Director — VIVUS LLC; Kishore Gadde, MD, Study Chair — Duke University
Locations (2):
- United States (2):
  - Research Site, Durham, North Carolina
  - Research Site, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at investigative sites in the US between November 2007 through January 2008
Groups:
- Placebo: Placebo
- PHEN 7.5 mg: 7.5 mg phentermine
- TPM 46 mg: 46 mg topiramate
- VI-0521 Mid: 7.5 mg/46 mg phentermine/topiramate
- PHEN 15 mg: 15 mg phentermine
- TPM 92 mg: 92 mg topiramate
- VI-0521 Top: 15 mg/92 mg phentermine/topiramate
Period: Overall Study
Arm/Group | Placebo | PHEN 7.5 mg | TPM 46 mg | VI-0521 Mid | PHEN 15 mg | TPM 92 mg | VI-0521 Top
Started | 109 | 109 | 108 | 107 | 108 | 107 | 108
Completed | 74 | 79 | 78 | 78 | 80 | 77 | 75
Not Completed | 35 | 30 | 30 | 29 | 28 | 30 | 33
Not completed — Lost to Follow-up | 14 | 14 | 12 | 6 | 9 | 8 | 9
Not completed — Adverse Event | 3 | 4 | 5 | 9 | 6 | 10 | 17
Not completed — Withdrawal by Subject | 11 | 6 | 5 | 7 | 8 | 5 | 4
Not completed — protocol non-compliance | 1 | 1 | 2 | 1 | 0 | 1 | 3
Not completed — Pregnancy | 1 | 0 | 1 | 2 | 1 | 2 | 0
Not completed — requirement for restricted medication | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Other | 5 | 5 | 3 | 4 | 4 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PHEN 7.5 mg | TPM 46 mg | VI-0521 Mid | PHEN 15 mg | TPM 92 mg | VI-0521 Top | Total
Number analyzed (Participants) | 109 | 109 | 108 | 107 | 108 | 107 | 108 | 756
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11.43) | 46.4 (11.57) | 46.9 (12.62) | 44.6 (11.07) | 45.7 (12.38) | 45.8 (11.21) | 44.6 (12.84) | 45.6 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 86 | 86 | 85 | 86 | 85 | 85 | 599
  Male | 23 | 23 | 22 | 22 | 22 | 22 | 23 | 157
Region of Enrollment [Number; unit: participants]
  United States | 109 | 109 | 108 | 107 | 108 | 107 | 108 | 756

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Loss From Baseline to Week 28
Description: Percent weight loss from baseline to Week 28 with last observation carried forward (LOCF)
Time Frame: baseline to 28 weeks
Population: Intent-to-treat Last-observation-carried-forward (ITT-LOCF)
Measure: Least Squares Mean (Standard Error); unit: percent weight loss
Arm/Group | Placebo | PHEN 7.5 mg | TPM 46 mg | VI-0521 Mid | PHEN 15 mg | TPM 92 mg | VI-0521 Top
Number analyzed (Participants) | 103 | 104 | 102 | 103 | 106 | 105 | 103
percent weight loss | 1.7 (0.61) | 5.5 (0.61) | 5.1 (0.61) | 8.5 (0.62) | 6.1 (0.61) | 6.4 (0.62) | 9.2 (0.61)
Statistical Analysis 1: Comparison: TPM 92 mg vs VI-0521 Top; With 100 subjects in each of the seven arms in this trial, the trial has more than 90% power to detect a difference of at least 3.1% between combination and monotherapy or placebo treatment assuming a standard deviation of 5.3% and a significance level of 0.05; Test type: Superiority or Other; p = 0.0009, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 2.76, 95% CI 2-sided [1.13 to 4.39], Standard Error of Mean 0.831
Statistical Analysis 2: Comparison: PHEN 15 mg vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 3.15, 95% CI 2-sided [1.53 to 4.77], Standard Error of Mean 0.825
Statistical Analysis 3: Comparison: Placebo vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 7.49, 95% CI 2-sided [5.86 to 9.12], Standard Error of Mean 0.830
Statistical Analysis 4: Comparison: TPM 46 mg vs VI-0521 Mid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 3.33, 95% CI 2-sided [1.69 to 4.96], Standard Error of Mean 0.832
Statistical Analysis 5: Comparison: PHEN 7.5 mg vs VI-0521 Mid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 3.01, 95% CI 2-sided [1.38 to 4.63], Standard Error of Mean 0.828
Statistical Analysis 6: Comparison: Placebo vs VI-0521 Mid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 6.75, 95% CI 2-sided [5.11 to 8.38], Standard Error of Mean 0.831

2. Primary Outcome: Percentage of Subjects With at Least 5% Weight Loss at Week 28 With LOCF
Time Frame: baseline to 28 weeks
Population: Intent-to-treat Last-observation-carried-forward (ITT-LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PHEN 7.5 mg | TPM 46 mg | VI-0521 Mid | PHEN 15 mg | TPM 92 mg | VI-0521 Top
Number analyzed (Participants) | 103 | 104 | 102 | 103 | 106 | 105 | 103
percentage of participants | 15.5 | 43.3 | 39.2 | 62.1 | 46.2 | 48.6 | 66.0
Statistical Analysis 1: Comparison: TPM 92 mg vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0140, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 2.028, 95% CI 2-sided [1.154 to 3.563], Standard Error of Mean 0.5832
Statistical Analysis 2: Comparison: PHEN 15 mg vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0046, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 2.246, 95% CI 2-sided [1.283 to 3.932], Standard Error of Mean 0.6418
Statistical Analysis 3: Comparison: Placebo vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 10.623, 95% CI 2-sided [5.424 to 20.81], Standard Error of Mean 3.6440
Statistical Analysis 4: Comparison: TPM 46 mg vs VI-0521 Mid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0011, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 2.568, 95% CI 2-sided [1.460 to 4.514], Standard Error of Mean 0.7391
Statistical Analysis 5: Comparison: PHEN 7.5 mg vs VI-0521 Mid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0066, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 2.166, 95% CI 2-sided [1.241 to 3.781], Standard Error of Mean 0.6158
Statistical Analysis 6: Comparison: Placebo vs VI-0521 Mid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 9.063, 95% CI 2-sided [4.650 to 17.66], Standard Error of Mean 3.0857

ADVERSE EVENTS:
Time Frame: AEs were collected from when written informed consent was provided through 28 days after the last dose of investigational product.
Description: Only subjects who received at least one dose of study drug were included in the safety analysis.
Arm/Group | Placebo | PHEN 7.5 mg | TPM 46 mg | VI-0521 Mid | PHEN 15 mg | TPM 92 mg | VI-0521 Top
Serious Adverse Events (participants affected / at risk) | 0/109 | 2/109 | 0/106 | 1/106 | 1/108 | 1/107 | 2/108
Other Adverse Events (participants affected / at risk) | 87/109 | 85/109 | 90/106 | 84/106 | 88/108 | 84/107 | 88/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=109) | PHEN 7.5 mg (N=109) | TPM 46 mg (N=106) | VI-0521 Mid (N=106) | PHEN 15 mg (N=108) | TPM 92 mg (N=107) | VI-0521 Top (N=108)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of ampulia of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic Mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cardiac arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=109) | PHEN 7.5 mg (N=109) | TPM 46 mg (N=106) | VI-0521 Mid (N=106) | PHEN 15 mg (N=108) | TPM 92 mg (N=107) | VI-0521 Top (N=108)
Bronchitis (Infections and infestations) | 3 | 2 | 2 | 6 | 3 | 2 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 12 | 9 | 13 | 14 | 9 | 14 | 14
Nasopharyngitis (Infections and infestations) | 11 | 6 | 10 | 3 | 10 | 9 | 11
Influenza (Infections and infestations) | 5 | 3 | 6 | 6 | 5 | 2 | 6
Sinusitis (Infections and infestations) | 6 | 3 | 5 | 2 | 8 | 5 | 4
Fatigue (General disorders) | 7 | 3 | 8 | 6 | 6 | 7 | 10
Irritability (General disorders) | 2 | 6 | 3 | 2 | 2 | 1 | 5
Insomnia (Psychiatric disorders) | 6 | 7 | 4 | 13 | 12 | 5 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 9 | 4 | 3 | 0 | 3 | 8
Vision blurred (Eye disorders) | 5 | 6 | 8 | 7 | 7 | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 4 | 1 | 6 | 1 | 9
Headache (Nervous system disorders) | 14 | 14 | 8 | 16 | 11 | 11 | 17
Paresthesia (Nervous system disorders) | 4 | 3 | 12 | 18 | 5 | 24 | 25
Dysgeusia (Nervous system disorders) | 0 | 1 | 7 | 9 | 1 | 2 | 16
Dizziness (Nervous system disorders) | 2 | 5 | 7 | 4 | 3 | 4 | 9
Disturbance in Attention (Nervous system disorders) | 1 | 1 | 2 | 7 | 1 | 4 | 4
Dry Mouth (Gastrointestinal disorders) | 0 | 8 | 7 | 14 | 13 | 7 | 20
Constipation (Gastrointestinal disorders) | 9 | 4 | 7 | 7 | 9 | 6 | 17
Nausea (Gastrointestinal disorders) | 5 | 5 | 8 | 9 | 6 | 5 | 8
Diarrhea (Gastrointestinal disorders) | 5 | 1 | 3 | 4 | 4 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.